CLINICAL TRIAL: NCT03523975
Title: Phase I/II Multi-site Study Evaluating the MTD, Safety and Efficacy of the Combination Venetoclax, Lenalidomide and Rituximab in Patients With Previously Untreated Mantle Cell Lymphoma
Brief Title: Venetoclax, Lenalidomide and Rituximab in Patients With Previously Untreated Mantle Cell Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19335; HUM00140979 (Other: University of Michigan)
Record Dates: First submitted 2018-04-26; First posted 2018-05-14 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — venetoclax; Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Venetoclax, Lenalidomide, Rituximab (Experimental): Rituximab 375 mg/m2 IV day 1, 8, 15, 22 of 1st cycle then on day 1 for cycles 2, 4, 6, 8, 10, 12 Lenalidomide 10 mg day 1-7 of and 15 mg day 8-14 cycle #1. 20 mg PO day day 15-21 of cycle #1 and days 1-21 cycles 2-12. Venetoclax PO days 8 - 28 cycles during cycle 1 only. Starting with ramp-up dose as follows (50 mg x 7 days then 100mg x 7 days then 200 mg x 7 days then 400 mg for remainder of therapy). Will be given days 1-28 at a dose of 400 mg cycle 2-12.
  Interventions: Drug: Venetoclax; Drug: Lenalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: Venetoclax — PO days 8 - 28 cycles during cycle 1 only. Starting with ramp-up dose as follows (50 mg x 7 days then 100mg x 7 days then 200 mg x 7 days then 400 mg for remainder of therapy). Will be given days 1-28 at a dose of 400 mg cycle 2-12.
Drug: Lenalidomide — 10 mg day 1-7 of and 15 mg day 8-14 cycle #1. 20 mg PO day day 15-21 of cycle #1 and days 1-21 cycles 2-12.
Drug: Rituximab — 375 mg/m2 IV day 1, 8, 15, 22 of 1st cycle then on day 1 for cycles 2, 4, 6, 8, 10, 12

SUMMARY:
The purpose of this study is to determine if giving an experimental drug called venetoclax in combination with lenalidomide and rituximab is safe and effective for treating people with Mantle Cell Lymphoma (MCL).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of mantle cell lymphoma (MCL) established by histologic assessment
* Laboratory, radiographic, physical exam findings and/or symptoms attributable to MCL
* ECOG Performance Status (Eastern Cooperative Oncology Group Performance Status: an attempt to quantify cancer patients' general well-being and activities of daily life. The score ranges from 0 to 5 where 0 is asymptomatic and 5 is death) less or equal to 2
* All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program.
* Men and Women of childbearing potential on appropriate contraception
* Adequate organ function
* Ability to understand and the willingness to sign a written informed consent.
* Ability to swallow oral capsules/tablets

Exclusion Criteria:

* Prior treatment for MCL with chemotherapy
* Pregnant or breastfeeding women
* Grade 2 or higher peripheral neuropathy
* Known history of CNS (Central Nervous System) or leptomeningeal by MCL prior to study enrollment
* Significant cardiovascular disease
* Any condition that might significantly impair drug absorption as determined by the investigator
* Uncontrolled active systemic fungal, bacterial, viral, or other infection, or intravenous anti-infective treatment within 2 weeks before first dose of study drug
* History of stroke or intracranial hemorrhage within 6 months of 1st dose of study drug
* Concurrent participation in another clinical trial
* Subject has received a moderate or strong CYP3A inhibitor or inducer within 1 week prior to treatment initiation.
* Psychiatric illness or social situations that would limit compliance with study requirements
* Subject has known positivity to HIV
* Active infection with Hepatitis B or C virus as determined by a detectable viral load on PCR.
* Prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or any other cancer from which the subject has been disease free for ≥ 2 years or which will not limit survival to< 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2018-12-24 (Actual); Primary Completion 2027-06-24 (Estimated); Study Completion 2027-06-24 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of the combination of lenalidomide, venetoclax and rituximab | 42 Days

SECONDARY OUTCOMES:
The proportion of patients with a Complete Response (CR) | Up to 4 Years
  Response will be assessed by the IRC (Immune-related Response Criteria) and the investigator on the basis of physical examinations and PET and CT scans using the Lugano 2014 criteria, taking into account results of bone marrow examinations for patients with bone marrow involvement at screening
The proportion of patients that respond to treatment | Up to 4 Years
  The proportion of patients who achieve either partial or complete response by PET, CT and marrow. Response will be assessed by the IRC and the investigator on the basis of physical examinations and PET and CT scans using the Lugano 2014 criteria, taking into account results of bone marrow examinations for patients with bone marrow involvement at screening

CONTACTS AND LOCATIONS:
Overall Officials: Tycel Phillips, M.D., Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical center, Duarte, California
  - University of Michigan, Ann Arbor, Michigan
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Phillips TJ, Bond D, Takiar R, Kump K, Kandarpa M, Boonstra P, Mayer TL, Nachar V, Wilcox RA, Carty SA, Karimi YH, Nikolovska-Coleska Z, Kaminski MS, Herrera AF, Maddocks K, Popplewell L, Danilov AV. Adding venetoclax to lenalidomide and rituximab is safe and effective in patients with untreated mantle cell lymphoma. Blood Adv. 2023 Aug 22;7(16):4518-4527. doi: 10.1182/bloodadvances.2023009992. PMID 37013954